CLINICAL TRIAL: NCT02427971
Title: A Comparison Between the Aysis® Cs2 (General Electrics) Ventilator in EtControl® Mode and the Perseus® A 500 (Dräger) in VaporView® Mode on Maniability and Consumption of Desflurane
Acronym: ConsoHalo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saint Antoine University Hospital (Other)
Responsible Party: Principal Investigator, Bonnot, MD, Saint Antoine University Hospital
Other Study IDs: 2014-A01476-41
Record Dates: First submitted 2015-04-15; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Anesthetics Agent; Consumption; Inhalation; Desflurane
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Perseus: Use of Perseus® A 500 with VaporView® mode that gives the evolution of inspired (Fi) and end-tidal (Fe) fractions of halogenated agents for 20 minutes based on the delivered fraction (Fd). FGF remains adjusted manually by the practitioner. This mode also makes it possible to maintain a low FGF (0.5 L/min)
- Aysis: Use of Aysis® Cs2 ventilator with automated control of end-tidal inhalation anesthetic concentration, EtControl® mode.

SUMMARY:
The Aysis® Cs2 ventilator offers an automated control of end-tidal inhalation anesthetic concentration, the EtControl® mode. A low Fresh Gas Flow (FGF) (0.5L/min) is kept during the maintenance of the anesthesia, decreasing the expensive consumption of halogenated agents.

The Perseus® A 500 offers a VaporView® mode that gives the evolution of inspired (Fi) and end-tidal (Fe) fractions of halogenated agents for 20 minutes based on the delivered fraction (Fd). FGF remains adjusted manually by the practitioner. This mode also makes it possible to maintain a low FGF (0.5 L/min), provided the halogen Fd is set to maintain a steady Fe curve.

The goal of this work was to compare the maniability of the intraoperative administered concentrations and the consumption of Desflurane between these 2 modalities of administration.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing a general anesthesia for intra abdominal surgery during more than one hour
* ASA 1or 2

Exclusion Criteria:

* contraindication to halogenated agent
* thoracic surgery
* no french speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA 1/2 adult patients undergoing a general anesthesia of more than one hour.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Consumption of Desflurane between these 2 modalities of administration. | Time of general anesthesia (1h minimum up to 12h)
  Des consumption was measured by micrometric weighing of the vaporizer before and after general anesthesia and a milliliter per min consumption was calculated

SECONDARY OUTCOMES:
Comparison of inspired (Fi) and end-tidal (Fe) fractions of halogenated evolution | Time of general anesthesia (1h minimum up to 12h)
Anesthesia depth monitoring by BIS | Time of general anesthesia (1h up to 12h)
Hemodynamic stability | Time of general anesthesia (1h minimum up to 12h)
  Number of cardiovascular event which required an intervention
  * Vasopressive drug
  * Antihypertensive drug
  * modification of the Desflurane end-tidal (Fe) fraction

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint-Antoine, Paris, France